CLINICAL TRIAL: NCT03512080
Title: National Institute of Health Research (NIHR) Global Health Research Group on Warfarin Anticoagulation in Patients with Cardiovascular Disease in Sub-Saharan Africa
Brief Title: Warfarin Anticoagulation in Patients in Sub-Saharan Africa
Acronym: War-PATH
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Professor Sir Munir Pirmohamed, David Weatherall Chair of Medicine and National Health Service (NHS) Chair of Pharmacogenetics, University of Liverpool
Other Study IDs: UoL001324
Record Dates: First submitted 2018-02-18; First posted 2018-04-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases
Keywords: Warfarin; Anticoagulation; Clinical Dosing Algorithm; Genetic Dosing Algorithm; International Normalised Ratio; Uganda; Cape Town; Cardiovascular Disease; Genome-wide Association Study; Stratified Medicine; Pharmacogenetics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stable International Normalised Ratio: Consenting adult patients with either venous thromboembolism (VTE), atrial fibrillation (AF) on warfarin with a target International Normalised Ratio (INR) (INR range 2-3) or valvular heart disease with a target INR (INR range 3-4).

SUMMARY:
This research programme aims to translate expertise in warfarin anticoagulation from resource-rich to low and middle income countries (LMIC)settings with the goal of improving patient health outcomes.

An observational study which will be used to develop warfarin dosing algorithms - the ultimate aim will be to ascertain whether these algorithms increase time in the therapeutic range, reduce bleeding and thrombotic risks, and clinic visits for International Normalised ratio (INR) monitoring. Two algorithms will be developed: the first will take into account clinical and geographical factors ("clinical algorithm"), while the second will also incorporate genetic factors in addition to the clinical and geographical factors ("genetic algorithm"). Patients will be recruited from sites in rural and urban Uganda, and in Cape Town, South Africa, to develop a clinical dosing algorithm. It is important to note that there is a wealth of literature data which will be used to define the clinical data that needs to be collected from these patients. To identify genetic factors in African patients, Genome-wide Association Study (GWAS) will be undertaken and any novel factors incorporated into the genetic algorithm - the percentage variation in warfarin dosing explained by the genetic algorithm will be compared with the clinical algorithm.

DETAILED DESCRIPTION:
This project focuses on an area unmet clinical need, oral anticoagulation, in patients with a variety of cardiovascular diseases. The investigators' ambition is to translate their internationally renowned expertise in warfarin anticoagulation into low and middle income country (LMIC) settings where it can significantly improve health. By working with policy makers, the investigators will provide the required evidence to allow national roll out of new practices, including the introduction of 1mg warfarin tablets as a quick win to improve dosing accuracy.

This National Institute of Health Research (NIHR) Global Research Group is a collaboration between the University of Liverpool and two low and middle income countries (LMICs), Uganda and South Africa. It will focus on a clinically important non-communicable disease area which requires the use of anticoagulation.

Anticoagulants, in particular warfarin, are used in these countries for the treatment of venous thromboembolism, valvular heart disease including rheumatic heart disease and prevention of strokes in patients with irregular heart rhythms (atrial fibrillation). Anticoagulation represents an unmet clinical need in Sub-Saharan Africa as patients either do not receive anticoagulation (because of difficulties in monitoring) or are poorly anticoagulated because of poor dosing guidelines. This results in potentially preventable morbidity and mortality which affects the poorer sectors of the population in particular. The investigators have extensive expertise in the United Kingdom and European Union of improving the use of warfarin through the development of novel dosing algorithms, which have now begun incorporating genetic factors.

By contrast, in the investigators' two collaborating partner countries, no locally validated warfarin dosing algorithms exist, even those which only take into account clinical factors. This results in haphazard dosing with the attendant risks of thrombotic or bleeding complications. In both countries, monitoring requires frequent clinic visits, incurring transport costs and missed work days. Patients are often co-infected with human immunodeficiency virus (HIV) and/or Tuberculosis, requiring multiple concomitant medicines which complicate warfarin dosing and dose adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adult patients with either venous thromboembolism (VTE), atrial fibrillation (AF) on warfarin with a target International Normalised Ratio (INR) (INR range 2-3) or valvular heart disease with a target INR (INR range 3-4).
2. On a stable maintenance dose for two consecutive clinic visits within the last six months, and the INR was in the therapeutic range at each of those visits.
3. Age over 18 years.
4. Self-reported Black African ethnicity.
5. Signed or witnessed written (witnessed thumbprint for illiterate participants) informed consent.

Exclusion Criteria:

1. Patient unwilling to take part.
2. Patient is, in the opinion of the investigator, not suitable to participate.
3. Pregnant women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Self-reported Black African ethnicity from Uganda and South Africa
Sampling Method: Non-Probability Sample
Enrollment: 681 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Identification of demographic, clinical and genetic factors in an African population that determine daily warfarin dosing requirements | 1 year
  Completion of an audit to evaluate the current quality of anticoagulant services in Cape Town and rural and urban Uganda taking into account the indications, anticoagulant clinic set-up and quality of anticoagulation control.
Development of a clinical algorithm taking into account patient factors, co-medications and underlying disease | 3 years
  Recruitment of patients currently on warfarin will be undertaken to identify clinical and other non-genetic factors associated with poor anticoagulation control to enable development of a warfarin clinical dosing algorithm. Data on patients' age, weight, height, gender, co-morbidities, co-medications, socio-economic factors, warfarin dose history and quality of anticoagulant control (International Normalised ratio (INR) measurement history) will be obtained for the algorithm development.
Development of a validated warfarin dosing algorithm taking into account both clinical and genetic factors | 3+ years
  Evaluation of genes specific to the local African populations in Uganda and South Africa that can impact on anticoagulation control will be carried out, resulting in the development of a novel genetic dosing algorithm. In order to identify ethnic specific genetic factors, the investigators will undertake a Genome-wide Association Study (GWAS) on these patients, and any novel genetic factors will be incorporated into an improved dosing algorithm which will be compared with the original algorithm in terms of its ability to predict therapeutic dose.

CONTACTS AND LOCATIONS:
Overall Officials: Munir Pirmohamed, Principal Investigator — University of Liverpool
Locations (2):
- University of Cape Town, Cape Town, South Africa
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adjusted-dose warfarin versus low-intensity, fixed-dose warfarin plus aspirin for high-risk patients with atrial fibrillation: Stroke Prevention in Atrial Fibrillation III randomised clinical trial. Lancet. 1996 Sep 7;348(9028):633-8. PMID 8782752
- [Background] Avery PJ, Jorgensen A, Hamberg AK, Wadelius M, Pirmohamed M, Kamali F; EU-PACT Study Group. A proposal for an individualized pharmacogenetics-based warfarin initiation dose regimen for patients commencing anticoagulation therapy. Clin Pharmacol Ther. 2011 Nov;90(5):701-6. doi: 10.1038/clpt.2011.186. Epub 2011 Sep 28. PMID 22012312
- [Background] Pirmohamed M. Warfarin: almost 60 years old and still causing problems. Br J Clin Pharmacol. 2006 Nov;62(5):509-11. doi: 10.1111/j.1365-2125.2006.02806.x. No abstract available. PMID 17061959
- [Background] Pirmohamed M, Burnside G, Eriksson N, Jorgensen AL, Toh CH, Nicholson T, Kesteven P, Christersson C, Wahlstrom B, Stafberg C, Zhang JE, Leathart JB, Kohnke H, Maitland-van der Zee AH, Williamson PR, Daly AK, Avery P, Kamali F, Wadelius M; EU-PACT Group. A randomized trial of genotype-guided dosing of warfarin. N Engl J Med. 2013 Dec 12;369(24):2294-303. doi: 10.1056/NEJMoa1311386. Epub 2013 Nov 19. PMID 24251363
- [Background] Pirmohamed M, James S, Meakin S, Green C, Scott AK, Walley TJ, Farrar K, Park BK, Breckenridge AM. Adverse drug reactions as cause of admission to hospital: prospective analysis of 18 820 patients. BMJ. 2004 Jul 3;329(7456):15-9. doi: 10.1136/bmj.329.7456.15. PMID 15231615
- [Background] Sekaggya C, Nalwanga D, Von Braun A, Nakijoba R, Kambugu A, Fehr J, Lamorde M, Castelnuovo B. Challenges in achieving a target international normalized ratio for deep vein thrombosis among HIV-infected patients with tuberculosis: a case series. BMC Hematol. 2016 Jun 4;16:16. doi: 10.1186/s12878-016-0056-6. eCollection 2016. PMID 27274846
- [Background] Wadelius M, Pirmohamed M. Pharmacogenetics of warfarin: current status and future challenges. Pharmacogenomics J. 2007 Apr;7(2):99-111. doi: 10.1038/sj.tpj.6500417. Epub 2006 Sep 19. PMID 16983400
- [Background] Cavallari LH, Perera MA. The future of warfarin pharmacogenetics in under-represented minority groups. Future Cardiol. 2012 Jul;8(4):563-76. doi: 10.2217/fca.12.31. PMID 22871196
- [Background] Mouton JP, Mehta U, Parrish AG, Wilson DP, Stewart A, Njuguna CW, Kramer N, Maartens G, Blockman M, Cohen K. Mortality from adverse drug reactions in adult medical inpatients at four hospitals in South Africa: a cross-sectional survey. Br J Clin Pharmacol. 2015 Oct;80(4):818-26. doi: 10.1111/bcp.12567. Epub 2015 Jul 6. PMID 25475751